CLINICAL TRIAL: NCT05164601
Title: A Multicenter, Prospective Cohort Study Evaluating the Prognosis of Patients with Acute Coronary Syndrome
Brief Title: Prognosis of Treated Acute Coronary Syndrome Patients: a Multicenter Study
Acronym: MPCS-ACS
Status: Completed | Type: Observational
Sponsor: Xiang Xie (Other)
Collaborators: Affiliated Traditional Chinese Medicine Hospital of Xinjiang Medical University (Unknown); The Third Affiliated Hospital of Jinzhou Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Xiang Xie, Head of Hypertension Department, Clinical Professor, Xinjiang Medical University
Organization: Xinjiang Medical University (Other)
Other Study IDs: xx20161107
Record Dates: First submitted 2018-11-07; First posted 2021-12-20 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Acute Myocardial Infarction; coronary heart disease; prognosis
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AMI Patients Cohort
  Interventions: Other: No Intervention - Observational Only

INTERVENTIONS:
Other: No Intervention - Observational Only — Clinical Follow-Up

SUMMARY:
The MPCS-ACS Study (Multicenter Prospective Cohort Study on Acute Coronary Syndrome) is a comprehensive, forward-looking research project designed to evaluate the prognostic outcomes of patients diagnosed with acute coronary syndrome (ACS) who declined coronary artery bypass grafting (CABG) and underwent percutaneous coronary intervention (PCI) instead. Leveraging a multicenter approach, the study aims to collect data from a diverse patient population, thereby enhancing the generalizability and clinical relevance of its findings.

Upon enrollment, detailed information is gathered, including demographic data, clinical history, and key biochemical markers. The study also documents the various medication regimens prescribed during hospitalization to assess their influence on patient outcomes. A key feature of MPCS-ACS is its rigorous follow-up protocol, which involves regularly monitoring patients after discharge to track recovery progress and the occurrence of any subsequent cardiovascular events.

This methodical approach is designed to generate valuable insights into the long-term prognosis of ACS patients treated with PCI, ultimately contributing to the refinement of therapeutic strategies and improving the standard of care across all participating centers.

DETAILED DESCRIPTION:
The Multicenter Acute Coronary Syndrome Prognosis Cohort Study (MPCS-ACS) is a comprehensive, longitudinal research initiative designed to evaluate the prognostic outcomes of patients diagnosed with acute coronary syndrome (ACS) across diverse healthcare settings. Conducted in collaboration with multiple hospitals, this study aims to collect and analyze data from ACS patients admitted between June 1, 2016, and May 31, 2021.

The study will gather an extensive range of variables, including therapeutic interventions, biochemical markers relevant to ACS management, as well as key demographic and clinical history data. By analyzing these factors, the study seeks to gain a deeper understanding of ACS treatment practices during the study period and assess their clinical efficacy.

A robust follow-up protocol is a cornerstone of MPCS-ACS, featuring routine evaluations conducted every six to twelve months after patient discharge. Follow-ups will incorporate both in-person visits and telecommunication to accommodate participants unable to return to the hospital. This dual approach is designed to maximize participant retention and ensure high-quality data collection, thereby enhancing the study's validity and impact.

Through its rigorous methodology and collaborative framework, the MPCS-ACS aims to identify key prognostic factors and outcomes for ACS patients. The ultimate goal is to inform the optimization of care strategies and elevate the standards of cardiovascular treatment across diverse healthcare systems.

ELIGIBILITY:
Inclusion Criteria

1. Men and women aged between 18 and 79 years.
2. Patients diagnosed with Acute Coronary Syndrome (ACS), including Unstable Angina (UA) and Acute Myocardial Infarction (AMI), based on typical clinical symptoms, changes in electrocardiographic (ECG) readings, and elevated cardiac biomarkers.
3. Patients who underwent coronary angiography confirming coronary artery stenosis and opted for PCI treatment instead of coronary artery bypass grafting (CABG).
4. Patients who are under long-term follow-up.

Exclusion Criteria

1. Patients with rheumatic heart disease, valvular heart disease, or congenital heart disease.
2. Patients with malignant tumors or hematologic diseases.
3. Patients with severe liver or kidney dysfunction or pulmonary heart disease.
4. Patients with a life expectancy of less than one year due to terminal illnesses such as advanced cancer or chronic kidney disease requiring dialysis.
5. Patients whose health is severely impacted by acute infections.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Coronary Syndrome
Sampling Method: Probability Sample
Enrollment: 22500 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Death | 10 years
  All-cause mortality, Cardiac mortality

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 10 years
  cardiac death, non-fatal myocardial infarction, significant aortic pathologies including aortic dissection and rupture of aortic aneurysms, episodes of unstable angina necessitating medical intervention, hospitalization for acute heart failure classified as Killip Class IV, and revascularization of the target vessel.
Major adverse cardiovascular and cerebrovascular events (MACCE） | 10 years
  cardiac death, non-fatal myocardial infarction, aortic events such as aortic dissection and aortic aneurysm rupture, episodes of unstable angina requiring medical intervention, hospitalization for acute heart failure assessed at Killip Class IV, target vessel revascularization, cerebrovascular events encompassing ischemic stroke, hemorrhagic stroke, transient ischemic attacks (TIAs) and subarachnoid hemorrhage.
revascularization of the target vesse | 10 years
  Revascularization of the target vessel was performed using percutaneous coronary intervention (PCI).
episodes of unstable angina necessitating medical intervention | 10 years
  Episodes of unstable angina requiring medical intervention were managed with urgent therapeutic measures.
hospitalization for acute heart failure classified as Killip Class IV | 10 years
  hospitalization for acute heart failure classified as Killip Class IV
non-fatal myocardial infarction | 10 years
  non-fatal myocardial infarction
cerebrovascular events | 10 years
  ischemic stroke, hemorrhagic stroke, transient ischemic attacks (TIAs) and subarachnoid hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Xie, PhD, Principal Investigator — Xinjiang Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medicial University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No